CLINICAL TRIAL: NCT05506007
Title: A Randomized, Open-label, Single Dose, Cross-over Clinical Trial to Compare the Safety, Tolerability, and Pharmacokinetic Properties of DA-5216 and DA-5216-R and to Evaluate the Food Effect on DA-5216 in Healthy Adult Subjects.
Brief Title: A Clinical Trial to Compare the Safety, Tolerability, and PK Properties of DA-5216 and DA-5216-R and to Evaluate the Food Effect on DA-5216.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA5216_BE_I
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- [Part A] DA-5216 (Experimental)
  Interventions: Drug: DA-5216
- [Part A] DA-5216-R (Experimental)
  Interventions: Drug: DA-5216-R
- [Part B] DA-5216(Fasting) (Experimental)
  Interventions: Drug: DA-5216
- [Part B] DA-5216(Fed) (Experimental)
  Interventions: Drug: DA-5216

INTERVENTIONS:
Drug: DA-5216 — During the cross-over [Part A], patients will be randomly assigned to receive one of the following treatment sequences:
  * Sequence I. Single dose of DA-5216-R(Fasting) on Day 1 followed by a single dose of DA-5216(Fasting) on Day 8.
  * Sequence II. Single dose of DA-5216(Fasting) on Day 1 followed by a single dose of DA-5216-R(Fasting) on Day 8.
  Arms: [Part A] DA-5216
Drug: DA-5216-R — During the cross-over [Part A], patients will be randomly assigned to receive one of the following treatment sequences:
  * Sequence I. Single dose of DA-5216-R(Fasting) on Day 1 followed by a single dose of DA-5216(Fasting) on Day 8.
  * Sequence II. Single dose of DA-5216(Fasting) on Day 1 followed by a single dose of DA-5216-R(Fasting) on Day 8.
  Arms: [Part A] DA-5216-R
Drug: DA-5216 — During the cross-over [Part B], patients will be randomly assigned to receive one of the following treatment sequences:
  * Sequence I. Single dose of DA-5216(Fasting) on Day 1 followed by a single dose of DA-5216(Fed) on Day 8.
  * Sequence II. Single dose of DA-5216(Fed) on Day 1 followed by a single dose of DA-5216(Fasting) on Day 8.
  Arms: [Part B] DA-5216(Fasting)
Drug: DA-5216 — During the cross-over [Part B], patients will be randomly assigned to receive one of the following treatment sequences:
  * Sequence I. Single dose of DA-5216(Fasting) on Day 1 followed by a single dose of DA-5216(Fed) on Day 8.
  * Sequence II. Single dose of DA-5216(Fed) on Day 1 followed by a single dose of DA-5216(Fasting) on Day 8.
  Arms: [Part B] DA-5216(Fed)

SUMMARY:
This is a randomized, open-label, single dose, 2-part, cross-over clinical trial to compare the safety, tolerability, and pharmacokinetic properties of DA-5216 and DA-5216-R and to evaluate the food effect on DA-5216 in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteer 19 years to 50 years
* Body weight in the range of 50.0kg and body mass index in the range of 18 to 27kg/m2
* Subject who are negative in pregnancy test or pregnant or Lactating women
* The subjects personally signed and dated informed consent document after informed of all patient aspects of the study, fully understanding and determined spontaneously to participate
* The subjects who are judged appropriate to participate this clinical trial according to the physical examination, routine laboratory examination and questionnaire

Exclusion Criteria:

* Subject with serious active hepatobiliary, respiratory, digestive, hematologic, endocrine(diabetes mellitus, aldosteronism), immunologic, cardiovascular(hypertension, angina, heart failure, myocardial infarction, etc.), neurologic, urologic, otorhinolaryngologic, musculoskeletal, psychological disease or history of such disease
* Subject with gastrointestinal disease (Crohn's disease, peptic ulcer, acute or chronic pancreatitis, etc.) or history of such disease/surgery (excluding simple appendic surgery, hernia surgery, hemorrhoid surgery).
* Subject who have galactose intolerance, Lapp lactase deficiency or glucose galactose malabsorption
* Subject who have had one or more of the following findings

  * AST, ALT > 1.5 times the upper limit
  * CPK > 2.5 times the upper limit
  * eGFR <60mL/min/1.73m2

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) PK parameter | 0~48hours
Area under the plasma concentration versus time curve (AUClast) PK parameter | 0~48hours

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hwan Lee, PhD, Principal Investigator — SNUH Clinical Pharmacololgy and Therapeutics
Locations (1):
- Seoul National University Hospital, Soeul, South Korea